CLINICAL TRIAL: NCT03649542
Title: The Effects of Fluidotherapy® Exercise on Wrist Fracture Rehabilitation Outcomes: A Pilot (Feasibility) Study
Brief Title: The Effects of Fluidotherapy® Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Collaborators: Summa Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUMMA IRB - FLUIDOTHERAPY
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Wrist Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pre/Post
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluidotherapy® plus exercises group (FLO) (Active Comparator): The Fluidotherapy® Unit and exercises group (FLO). They were required to complete wrist exercises in Fluidotherapy® Unit box for 15 minutes with the following exercises finger abduction/adduction, finger flexion/extension, forearm supination/pronation, wrist flexion/extension, and wrist radial deviation/ulnar deviation. Each patient performed two sets of fifteen repetitions for each exercise, totaling 15-minutes.
  Interventions: Other: Fluidotherapy plus exercise
- Exercises only group (EX) (No Intervention): They were required to complete wrist exercises in the air for 15 minutes, including abduction/adduction, finger flexion/extension, forearm supination/pronation, wrist flexion/extension, and wrist radial deviation/ulnar deviation. Each patient performed two sets of fifteen repetitions for each exercise, totaling 15-minutes.

INTERVENTIONS:
Other: Fluidotherapy plus exercise — The Fluidotherapy® unit (ULTRA 115: Henley International, Sugar Land, Texas) is a high intensity heat modality consisting of a dry whirlpool of finely divided solid particles suspended in a heated air stream. A certified technician The cleaned the Fluidotherapy® unit per the user manual.
  Other Names: Exercise Only
  Arms: Fluidotherapy® plus exercises group (FLO)

SUMMARY:
BACKGROUND: Wrist fractures are a common upper extremity injury treated by hand therapists. Currently, there is a dearth of published literature supporting the use Fluidotherapy® to improve pain and range of motion (ROM) in wrist fracture patients. \OBJECTIVE: This pilot study was conducted to determine the effects of one 15-minute bout of performing active range of motion (AROM) exercises in Fluidotherapy® (EXFT) versus AROM exercises (EX) alone on pain levels and AROM in wrist fracture subjects. METHODS: Eight subjects diagnosed with a wrist fracture (distal radius fracture, distal radius/ulna fractures, or distal ulna fracture) and referred to outpatient rehabilitation/occupational therapy were recruited upon his/her initial therapy evaluation. RESULTS: There were no significant differences between EX and EXFT groups in all outcome variables except for self-reported numeric pain scores (p=0.03*) and a trend towards significance in pronation AROM (p=0.06**). Even with a small sample size (n=8) there were significant differences in self-reported pain between the two groups. CONCLUSION: This study confirms that even after one 15-minute bout of AROM exercises in Fluidotherapy® treatment, patients report improved pain tolerance and may be useful in pain management techniques after a wrist fracture.

DETAILED DESCRIPTION:
BACKGROUND: Wrist fractures are a common upper extremity injury treated by hand therapists. Fluidotherapy® is a high intensity heat modality consisting of a dry whirlpool of finely divided solid particles suspended in a heated air stream, the mixture having the properties of a liquid. Currently, there is a dearth of published literature supporting the use Fluidotherapy® to improve pain and range of motion (ROM) in wrist fracture patients. More importantly, there is no evidence for the reduction of perceived wrist pain or improved ROM after only one 15-minute bout of Fluidotherapy®. OBJECTIVE: This pilot study was conducted to determine the effects of one 15-minute bout of performing active range of motion (AROM) exercises in Fluidotherapy® (EXFT) versus AROM exercises (EX) alone on pain levels and AROM in wrist fracture subjects. METHODS: Eight subjects diagnosed with a wrist fracture (distal radius fracture, distal radius/ulna fractures, or distal ulna fracture) and referred to outpatient rehabilitation/occupational therapy were recruited upon his/her initial therapy evaluation. Patients with closed reductions, open reductions, internal fixation, and/or external fixation were included as well. Subjects were randomly assigned to either the EXFT group or the EX group. A numeric pain scale (0-10) was used to assess perceived pain and AROM measurements using a goniometer were taken for pronation, supination, flexion, extension, radial deviation, and ulnar deviation immediately prior to intervention and after intervention. RESULTS: EX Group Pre-Treatment results: Pain 4.0 (± 1.82); Supination AROM 75.5 (± 10.90); Pronation AROM 75 (± 7.02); Flexion AROM 34.5 (± 9.88); Extension AROM 43.5 (± 8.96); Radial Deviation AROM 18.75 (± 9.43); Ulnar Deviation AROM 23.5 (± 4.36); Exercise in Fluidotherapy® Group Pre-Treatment results: Pain 2.5 (± 2.08); Supination AROM 65 (± 18.70); Pronation AROM 81.25 (± 6.29); Flexion AROM 40.25 (± 17.23); Extension AROM 38.5 (± 12.07); Radial Deviation AROM 21.25 (± 10.31); Ulnar Deviation AROM 26.25 (± 12.5); EX Group Post-Treatment results: Pain 4.5 (± 2.52); Supination AROM 81.75 (± 9.18); Pronation AROM 79 (± 3.46); Flexion AROM 36.25 (± 9.84); Extension AROM 50.5 (± 15.42); Radial Deviation AROM 21.5 (± 9.94); Ulnar Deviation AROM 23.75 (± 5.19); Exercise in Fluidotherapy® Group Pre-Treatment results: Pain 0.75 (± 0.98); Supination AROM 72.5 (± 14.43); Pronation AROM 86.25 (± 4.79); Flexion AROM 47.5 (± 15.54); Extension AROM 51.25 (± 8.54); Radial Deviation AROM 25.5 (± 12.80); Ulnar Deviation AROM 29 (± 8.41); There were no significant differences between EX and EXFT groups in all outcome variables except for self-reported numeric pain scores (p=0.03*) and a trend towards significance in pronation AROM (p=0.06**). Even with a small sample size (n=8) there were significant differences in self-reported pain between the two groups. CONCLUSION: The application of heat, massage, sensory stimulation, levitation, and pressure oscillations seem to provide patients pain relief and improvements in range of motion after AROM exercises in Fluidotherapy®. This study confirms that even after one 15-minute bout of AROM exercises in Fluidotherapy® treatment, patients report improved pain tolerance and may be useful in pain management techniques after a wrist fracture.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be referred to outpatient rehabilitation at St. Thomas Hospital, Akron, Ohio.
* Patients diagnosed with a wrist fracture will include those patients with distal radius fractures, distal radius/ulna fractures, and distal ulna fractures. Patients who have had closed reductions, open reductions, internal fixation, and/or external fixation will all be included.
* Patients will be recruited for this study if they have been cleared by the referring physician on the order to safely begin wristrange of motion.

Exclusion Criteria:

* Have open wounds
* Have Hepatitis
* Currently have chicken pox or shingles
* Have other serious fractures in the arm
* Have blood circulation problems in the arms or legs
* Do not have a physician referral to outpatient rehab
* Fractured wrist less than 6-weeks old as of evaluation day
* Fractured wrist over a year ago
* Under the age of 18 and over the age of 85 years at the time of participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-07-27 (Actual); Primary Completion 2014-01-13 (Actual); Study Completion 2014-01-13 (Actual)

PRIMARY OUTCOMES:
active range of motion (AROM) | 15 minutes after
  Using a goniometer, Scale and measured the patient's supination, pronation, wrist flexion and extension, wrist radial deviation, and wrist ulnar deviation.

IPD SHARING:
Plan to Share IPD: No